CLINICAL TRIAL: NCT05427201
Title: Integrated Repetitive Transcranial Magnetic Stimulation and Acceptance and Commitment Therapy for Veterans With Chronic Pain and Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation and Acceptance and Commitment Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4090-P; RX004090 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Depression
Keywords: Chronic pain; Depression; Repetitive transcranial magnetic stimulation; Acceptance and commitment therapy
MeSH Terms: conditions — Chronic Pain; Depression | interventions — Transcranial Magnetic Stimulation; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DLPFC-rTMS + ACT (Experimental): Active DLPFC-rTMS with ACT treatment
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Acceptance and Commitment Therapy
- Sham-rTMS + ACT (Active Comparator): Sham delivered rTMS with ACT treatment
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive brain stimulation technique designed to alter network function
  Other Names: rTMS
  Arms: DLPFC-rTMS + ACT
Behavioral: Acceptance and Commitment Therapy — ACT is a mindfulness-based cognitive behavioral intervention that has demonstrated efficacy for chronic pain.
  Other Names: ACT

SUMMARY:
Veterans with comorbid chronic pain and depression are highly prevalent, have poor functional status and low quality of life, are at increased risk of suicide and lack access to effective treatments. To address this problem, the proposed research will examine the feasibility of a novel approach that integrates repetitive Transcranial Magnetic Stimulation and Acceptance and Commitment Therapy with the overall goal of maximizing functional improvement in Veterans with chronic pain and depression. This is an important first-step in preparation for a future randomized efficacy trial. The investigators will also include two cognitive control tasks with concurrent electroencephalography to explore as a potential objective indicator of treatment response. This application addresses a critical need within the Veterans Health Administration and is closely aligned with the focus area of developing suicide prevention treatments that influence participation in life roles.

DETAILED DESCRIPTION:
Comorbid depression is highly prevalent in Veterans with chronic pain and contributes to greater pain severity, functional impairment, and suicide risk relative to those with chronic pain alone. Despite the well-known association between chronic pain and depression, current treatments fall short of producing meaningful improvements in function and quality of life in this population. In this application, the investigators propose to address this problem by a novel intervention that combines repetitive Transcranial Magnetic Stimulation (rTMS) and Acceptance and Commitment Therapy (ACT).

ACT is an evidence-based psychosocial intervention that improves function in Veterans with chronic pain. However, similar to the broader literature, comorbid depression significantly limits the efficacy of ACT, which may be directly related to dysfunctional brain circuits that maintain depression. rTMS is a non-invasive brain stimulation intervention that is FDA-cleared for the treatment of depression. The most commonly targeted stimulation area is the left dorsolateral prefrontal cortex (DLFPC), a prefrontal brain region involved in cognitive control and emotion regulation. rTMS over the left DLPFC has also been used to reduce pain intensity in patients with chronic pain, as the DLPFC is implicated in the affective processing of painful stimuli. Importantly, while rTMS has been shown to reduce depression severity and pain intensity, it does not directly address function. Thus, the proposed research will integrate rTMS and ACT with the goal of maximizing functional improvement in Veterans with chronic pain and depression.

The purpose of this application is to examine the feasibility of a future randomized efficacy trial. A total of 24 Veterans with chronic pain and depression will be randomized into DLPFC-rTMS + ACT or sham-rTMS + ACT conditions. Multiple metrics of feasibility will be assessed, including general interest in the study, willingness to participate, enrollment, retention, drop-out, number of adverse events, and participant blindness to condition, as well as ratings of credibility, expectation, and treatment satisfaction. The investigators will also estimate the preliminary impact of DLPFC-rTMS + ACT and sham-rTMS + ACT on function as measured by reductions in pain interference (primary clinical outcome). The intent of preliminary analyses is to obtain an additional indicator for a future large-scale trial, not to verify group differences. Further, the investigators will include two cognitive control tasks, the Emotion Distractor and Attention-to-Breath tasks, with concurrent EEG recording as a potential objective indicator of treatment response. The study team has previously demonstrated the association between depression severity and DLPFC activity on these tasks. In the proposed study, the investigators will explore the associations between treatment-related change in DLPFC activity and treatment outcomes.

Veterans with chronic pain and depression do not have access to effective treatments. To address this need, the investigators seek to examine the feasibility of a novel approach by integrating a somatic and a psychosocial intervention. The investigator's scientific premise is that rTMS over the left DLPFC will remediate hypofunction of prefrontal brain circuits that is necessary to maximize the impact of ACT on function in Veterans with chronic pain and depression. Findings from the proposed research have the potential of substantially increasing the physical and psychosocial functioning of Veterans with chronic pain and depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chronic, non-terminal pain condition (pain most days for at least 6 months)
* Average pain intensity and interference with enjoyment of life and/or general activity rated > 4/10 over the past week, as measured by the PEG
* Meet clinical criteria for major depression via DSM5 criteria, as assessed by the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Serious or unstable medical illness (e.g., cardiovascular disease)
* Lifetime history of psychotic disorder, bipolar disorder, obsessive-compulsive disorder
* Active substance abuse or psychosocial instability (e.g., homelessness) that could compromise study participation
* Changes to professionally delivered pain or mood treatment (e.g., no discontinuation of a treatment; no increasing the dose of medication) one month preceding the baseline assessment
* Significant neurologic disorder, increased risk of seizure for any reason or family/personal history of seizure
* Contraindications to rTMS treatment as outlined by the Safety of TMS Consensus group, which includes implanted metallic objects above the neck, implanted electrical devices (pacemakers/spinal cord stimulators), and pregnancy
* Prior trial of rTMS for any condition and/or lack of responsiveness to electroconvulsive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference change | Baseline, weekly during ACT intervention, 9 weeks
  The PROMIS Pain Interference questionnaire consists of 8-items that assess the degree to which pain interferes with various aspects of life, including mobility, social activity, and mood. Items are scored on a 1 ("Not at all") to 5 ("Very much") scale with a range of 8 - 40. Higher scores indicate greater pain interference.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) change | Baseline, weekly during ACT intervention, 9 weeks
  The PHQ-9 is a widely used measure of depressive symptoms. Items are scored on a 0 ("not at all") to 3 ("Nearly every day") scale with a range of 0 - 27. Higher scores indicate greater depression severity.
PROMIS Pain Intensity change | Baseline, weekly during ACT intervention, 9 weeks
  The PROMIS Pain Intensity questionnaire consists of 3 items assessing worst and average pain over the past week, as well as current pain. Items are scored on a 1 ("No pain") to 5 ("Very severe") scale with a range of 3 - 15. Higher scores indicate greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Herbert, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A data repository will be created upon completion of the study. Data obtained in this study that has scientific value to other qualified researchers will made available upon request. Interested researches will be able to access de-identified data through a Data Use Agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Indefinitely
Access Criteria: January, 2025

DOCUMENTS (1):
  • Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05427201/ICF_000.pdf